CLINICAL TRIAL: NCT03056443
Title: Initiation of CPAP for Newly Diagnosed OSA in Hospitalized Heart Failure Patients: A Randomized Clinical Trial
Brief Title: Initiation of CPAP for Newly Diagnosed OSA in Hospitalized Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Robert Stansbury, MD, Associate Professor, Sleep Medicine Fellowship Program Director, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WVU02HSC16
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Sleep Apnea, Obstructive; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Heart Failure | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Positive Airway Pressure-CPAP (Experimental): CPAP education and discharge with auto-adjusting Continuous Positive Airway Pressure (CPAP) in addition to usual standards of clinical care for heart failure.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Standard of Care (No Intervention): CPAP initiation per standard of care based on approval by insurance company and DME company with management as per usual standards of clinical care for heart failure.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — The auto-CPAP group will be scheduled for follow-up with a phone call at 2 - 3 weeks post discharge, then in sleep medicine clinic at 1 month (+2 weeks) and 6 months (+2 weeks) to assess their progress on CPAP.
  Arms: Continuous Positive Airway Pressure-CPAP

SUMMARY:
The study aimed to examine the effect of Continuous Positive Airway Pressure (CPAP) initiation for newly diagnosed obstructive sleep apnea (OSA) in hospitalized heart failure patients on reducing 30-day hospital readmission rate through a clinical trial.

DETAILED DESCRIPTION:
Following consent adult patients hospitalized with a medical history of heart failure and meeting study eligibility criteria will be screened for obstructive sleep apnea using the Ohio Sleep Medicine Institute Preoperative Questionnaire.

If the probability of sleep apnea is high (Sleep apnea clinical Score >15) then participants will complete the Epworth Daytime Sleepiness scale and the Minnesota Living with HeartFailure questionnaire. The patient will then be evaluated by the sleep medicine team with a portable polysomnography monitor which has been shown to be equivalent to standard in-laboratory polysomnography. All participants with apnea-hypopnea index (AHI) ≥ 5events/h in whom sleep disordered breathing is confirmed by sleep medicine physician will be eligible for randomization.

Participants will be randomized into an auto-adjusting Continuous Positive Airway Pressure (CPAP) group or standard of care (control) group.

CPAP Arm (Intervention): CPAP education and discharge with auto-adjusting Continuous Positive Airway Pressure (CPAP) in addition to usual standards of clinical care for heart failure. The auto-CPAP group will be scheduled for follow-up with a phone call at 2 - 3 weeks post discharge, then in sleep medicine clinic at 1 month (+2 weeks) and 6 months (+2 weeks) to assess their progress on CPAP.

Standard of Care Arm (Comparator): CPAP initiation per standard of care based on approval by insurance company and DME company with management as per usual standards of clinical care for heart failure. This group will be scheduled for follow-up with a phone call at 2- 3 weeks post discharge and then in sleep medicine clinic at 1 month (+2 weeks) and 6 months (+2 weeks) to assess their progress.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized having a documented history of heart failure
* Anticipated hospitalization of more than 24 hours
* Subject has obtained a score of > 15 on the Ohio Sleep Medicine Institute Preoperative questionnaire.
* Subject has an apnea-hypopneas index (AHI) of > 5/h as confirmed by sleep medicine physician

Exclusion Criteria:

* The presence of any conditions that the investigator feels will interfere with the use of CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stansbury, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stansbury R, Abdelfattah M, Chan J, Mittal A, Alqahtani F, Sharma S. Hospital screening for obstructive sleep apnea in patients admitted to a rural, tertiary care academic hospital with heart failure. Hosp Pract (1995). 2020 Dec;48(5):266-271. doi: 10.1080/21548331.2020.1799601. Epub 2020 Aug 4. PMID 32715796

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No subjects enrolled in arm for no intervention: standard of care.
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure-CPAP
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No subjects enrolled into arm "No intervention: Standard of Care"
Arm/Group | Continuous Positive Airway Pressure-CPAP
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 57.9 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Epworth Sleepiness Scale Score [Median (Full Range); unit: units on a scale] — 0-5 Lower Normal Daytime Sleepiness 6-10 Higher Normal Daytime Sleepiness 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness 16-24 Severe Excessive Daytime Sleepiness
  units on a scale | 15.4 [5 to 24]
Minnesota Heart Failure Questionnaire [Median (Full Range); unit: Score on a scale] — Minnesota Living with Heart Failure Questionnaire (MLHFQ) will be used to determine the disease-specific quality of life. It has 21 items in physical, emotional and socioeconomic dimensions; each item scored from 0 to 5 [For each question the answer may vary from 0 (no), 1 (very little) to 5 (very much)] provides a total score between 0 to 105: the higher the score, the lower quality of life.
  Score on a scale | 71.7 [0 to 105]
Distance Lived from Sleep Center [Median (Full Range); unit: Miles] | 55.7 [6 to 183]
Apnea Hypopnea Index [Median (Full Range); unit: events/hour] | 16.4 [5.6 to 56.7]

OUTCOME MEASURES:

1. Primary Outcome: All-cause Hospital Readmission Within 30 Days of Hospital Discharge.
Description: Thirty-day hospital readmission will be defined as a hospitalization or visit to the emergency department (ED) for a cardiac cause > 48 h after discharge. A readmission will be defined as a hospitalization for any reason within 30 days after discharge, and only the first readmission will be counted in case of multiple readmission in the 30-day period.
Time Frame: From hospital discharge to any hospitalization readmission within 30 days from discharge
Population: No subjects enrolled into arm "No intervention: Standard of Care"
Measure: Number; unit: readmissions
Arm/Group | Continuous Positive Airway Pressure-CPAP
Number analyzed (Participants) | 13
readmissions | 3

ADVERSE EVENTS:
Time Frame: 6 months + 2 weeks
Description: No subjects were enrolled into arm "No intervention: Standard of Care"
Arm/Group | Continuous Positive Airway Pressure-CPAP
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Positive Airway Pressure-CPAP (N=13)
Readmission (General disorders) | 1 (2)
Readmission (General disorders) | 1 (1) — Morphine Overdose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03056443/Prot_SAP_000.pdf